CLINICAL TRIAL: NCT01316458
Title: An Open-label, Multicenter, Phase II Study to Evaluate the Ability of Glivec® (Imatinib, Formerly Known as STI571) to Produce a Biochemical Response in Patients With Rising PSA Following Radical Prostatectomy
Brief Title: Glivec in Prostate Cancer Patients With Rising PSA Following Radical Prostectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571BDE15
Record Dates: First submitted 2011-03-14; First posted 2011-03-16 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2011-03

CONDITIONS: Prostatic Neoplasm; Genital Neoplasms, Male; Neoplasms, Abdominal; Urogenital Neoplasms; Genital Diseases, Male; Prostatic Diseases; Antineoplastic Agents; Imatinib
Keywords: Prostate cancer,; radical prostatectomy,; PSA rise
MeSH Terms: conditions — Prostatic Neoplasms; Genital Neoplasms, Male; Abdominal Neoplasms; Urogenital Neoplasms; Genital Diseases, Male; Prostatic Diseases | interventions — Imatinib Mesylate

ARMS (1):
- imatinib mesylate (Experimental)
  Interventions: Drug: STI571 (Glivec®)

INTERVENTIONS:
Drug: STI571 (Glivec®)
  Other Names: Glivec

SUMMARY:
To investigate the ability of 600 mg of Glivec®, given once daily by mouth to patients with rising PSA following radical prostatectomy, to produce a sustained biochemical response during the first 6 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* who are 18 years of age or older.
* who have undergone radical prostatectomy within 2 years prior to PSA progression .
* exhibiting two consecutive rises in PSA levels relative to a previous reference value, separated by 14 days.

The first measurement must occur 14 days after the reference value und must be at least 20% above the reference value. The reference value must be at least 0.4 ng/ml. The second confirmatory measurement taken 14 days after the first measurement must be greater than the first measurement.

* with a Karnofsky Performance Score (KPS) greater than or equal to 90 (Appendix 5).
* with the following hematologic lab values: ANC greater than or equal to 1500/mm3, Hgb greater than or equal to 10g/dL, PLT greater than or equal to 100x109/L.
* with the following biochemistry lab values: total bilirubin < 1.5 ULN, SGOT, SGPT less than or equal to 2.5 ULN, serum creatinine less than or equal to 1.5 ULN.
* willing to employ an effective barrier method of contraception during the study duration and for 3 months following discontinuation of study drug (for patients of reproductive potential).
* with a life expectancy of > 6 months.
* who have provided written informed consent pursuant to local regulatory requirements prior to initiation of any study procedure.

with a Gleason Score > 6 in the prostatectomy specimen

Exclusion Criteria:

* with a history of another malignancy within 5 years prior to study entry, except curatively treated non-melanotic skin cancer, unless written approval is obtained by the sponsor.
* with prior hormonal therapy
* who require therapy with warfarin or analgesics of the morphine class or higher (see Section 3.4.4).
* with a known diagnosis of HIV, hepatitis B, or hepatitis C infection.
* who have had a major surgery within 2 weeks prior to study entry.
* with severe, unstable, or uncontrolled medical disease which would confound diagnoses or evaluations required by the protocol, including severe cardiac insufficiency (NYHA III or IV, see Appendix 2), uncontrolled diabetes, chronic hepatic or renal disease, and active uncontrolled infection.
* with a history of noncompliance to medical regimens or inability or unwillingness to return for all scheduled visits.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2003-06; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
investigate the ability of 600 mg of Glivec®, given once daily by mouth to patients with rising PSA following radical prostatectomy, to produce a sustained biochemical response during the first 6 months of treatment. | 2 - 4 weeks

SECONDARY OUTCOMES:
investigate the time to sustained biochemical response under the treatment of Glivec® in this patient population | continuous
investigate duration of biochemical sustained response under the treatment with Glivec® in this patient population. | continuous
To assess the response rates: number of patients with complete, partial and minor biochemical response and stable PSA | continuous
To assess the time to clinical progression of this patient population treated with Glivec® at this dose and schedule. | continuous
To descriptively characterize the safety and tolerability of Glivec® administered at this dose and schedule to this patient population. | continuous

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- Germany (13):
  - Novartis Investigative Site, Aachen
  - Novarts Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Borken
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Fürth
  - Novartis Investigative Site, Gardelegen
  - Novarts Investigative Site, Hamburg
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Wesel
  - Novartis Investigative Site, Wuppertal